CLINICAL TRIAL: NCT06422559
Title: Accelerated Intermittent Theta Burst Stimulation in Unipolar Versus Bipolar Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.22.12.731
Record Dates: First submitted 2024-04-23; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants with unipolar depression (Experimental): Participants with Unipolar depression will receive 30 sessions of TMS.10 sessions a week for 3 weeks
  Interventions: Device: Transmagnetic stimulation; Device: TMS
- Participants with bipolar depression (Experimental): Participants with bipolar depression will receive 30 sessions of TMS.10 sessions a week for 3 weeks
  Interventions: Device: Transmagnetic stimulation; Device: TMS

INTERVENTIONS:
Device: Transmagnetic stimulation — Stimulatory TMS protocol using MagVenture MagPro R30 stimulator with the Cool-B65 coil
Device: TMS — Stimulatory TMS protocol using MagVenture MagPro R30 stimulator with the Cool-B65 coil

SUMMARY:
The goal of this interventional study is to learn if accelerated Intermittent Theta Burst Stimulation can improve symptoms of 30 participants with Unipolar depression in higher manner than symptoms of 30 participants with bipolar depression

DETAILED DESCRIPTION:
We will apply stimulatory TMS protocol for participants with Unipolar depression and participants with bipolar depression using MagVenture MagPro R30 stimulator with the Cool-B65 coil

ELIGIBILITY:
Inclusion Criteria:

* Age:18_65 years
* Sex:male and female
* Patients with Unipolar depression and bipolar depression diagnosis confirmed by SCID according to DSM5
* No pharmacological change in the last 4 weeks before the beginning of the stimulantion cycle
* Pharmacological resistance

Exclusion Criteria:

* Patients complaining of psychosis.Substance Use Disorder.current suicidal ideation.major medical and neurological disorder
* Patients complaining of epilepsy
* pregnancy and breastfeeding
* peacemaker spinal or bladder stimulator
* History of skull surgery and trauma
* presence of metallic foreign body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of severity of manic symptoms before and after treatment | One year for completion of the study
  We will use Young Mania Rating Scale._Young Mania Rating Scale:assess severity of manic symptoms, clinician rated,<=12(remission)13_19(minimal symptoms)20_25(mild mania)26_37(moderate mania)38_60 severe mania
Comparison of the severity of the patient's illness at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis. | One year for completion of the study
  We will use Clinical Global Impression Severity Scale._Clinical Global Impression Severity Scale:rate the severity of the patient's illness at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis,1 normal not at all ill,2 borderline mentally ill,3 mildly ill,4 moderately ill,5 markedly ill,6 severely ill,7 extremely ill
Comparison of severity and impact of insomnia before and after treatment | One year for completion of the study
  We will use Insomnia Severity Index scale._Insomnia Severity Index:assess the nature, severity and impact of insomnia,0_7(absence insomnia) 8_14(subthreshold insomnia)15_21(moderate insomnia)22_28(severe insomnia)
Comparison of depressive symptoms before and after treatment | One year for completion of the study
  We will use Hamilton Depression Rating Scale._Hamilton Depression Rating Scale:assess the severity of depressive symptoms, clinician rated,0_7(normal range)8_16(mild severity)17_23(moderate severity)>23(severe depression)

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. El-boraie, Study Chair — Professor; Ibrahim H. Rashed, Study Director — Assistant professor; Hassan M. Sonbol, Study Director — Lecturer
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang J, Chu Y, Ren Y, Li C, Wang Y, Chu XP. Maintenance treatment of transcranial magnetic stimulation (TMS) for treatment-resistant depression patients responding to acute TMS treatment. Int J Physiol Pathophysiol Pharmacol. 2020 Oct 15;12(5):128-133. eCollection 2020. PMID 33224435
- See also: PMC 7675193 — https://pubmed.ncbi.nlm.nih.gov/33224435/